CLINICAL TRIAL: NCT00358852
Title: Scale Validation of Prediction of Relapse and Rehospitalization Short Term in Patients With Schizophrenia
Brief Title: Scale Validation Study for Prediction of Relapse and Short Term Rehospitalization in Patients With Schizophrenia
Acronym: PRE-COG
Status: Completed | Type: Observational
Sponsor: Janssen-Cilag, S.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR011989; RISSCH4075 (Other: Janssen-Cilag S.A., Spain); NCT01991496 (obsolete NCT alias)
Record Dates: First submitted 2006-07-28; First posted 2006-08-01 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-03

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Mental disorder; Schizoaffective disorder; Schizophreniform disorder; Epidemiological study; Scale validation; Relapse; Short Term Hospitalization; PRE-COG; RISSCH4075
MeSH Terms: conditions — Schizophrenia; Mental Disorders; Psychotic Disorders; Recurrence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with Schizophrenia
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is an observational study. The data will be collected of patients suffering from schizophrenia and schizoaffective disorder / schizophreniform.

SUMMARY:
The purpose of this study is to establish and validate a scale/model that can be used to evaluate the duration of time and factors between short term hospital treatment and subsequent relapse periods in patients with schizoaffective/schizophreniform disorders.

DETAILED DESCRIPTION:
This is an epidemiological (study of the distribution and determinants of health-related states or events in defined population), multicenter (study conducted at multiple sites), observational (study in which patients are observed), cross-sectional (observation of all patients at one specific point in time), prospective (in which the patients are first identified and then followed forward as time passes) study. The sources of information in the study are units medical short stay psychiatric hospitalization or the acute care of the whole country, and clinical data of the patient at discharge. No intervention will be provided in this study. The general data (age range, gender, highest level of educational attainment, level of family support, substance abuse, events stressors, type of schizophrenia according to DSM-IV criteria [Diagnostic and Statistical Manual fourth], etc) of approximately 2000 schizophrenia and schizoaffective disorder / schizophreniform patients will be collected in this study. No special tests will be done during the study. The study will collect patients' data in electronic data collection workbook and model validation will be used at 6 and 12 months to confirm no relapse / hospitalization. The study observation period corresponds to the 3 years preceding the current relapse and current income (current hospitalization period) and 12 months after admission.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Schizophrenia or Schizoaffective disorder of more than 2 years evolution and who find themselves admitted in a Short-Term Psychiatric Hospitalization Unit or Acute Unit

Exclusion Criteria:

* Other patients with a psychiatric pathology different to schizophrenia, schizoaffective/schizophreniform disorders
* Patients with schizophrenia or schizoaffective/schizophreniform disorders of 2 years, or less evolution
* Pregnant, lactating, or planning to become pregnant within the next 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with schizophrenia, schizoaffective / schizophreniform more than 2 years of evolution and who are admitted to inpatient psychiatric units for short stay acute care setting.
Sampling Method: Non-Probability Sample
Enrollment: 2339 (Actual)
Dates: Start 2006-08; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Time to short-term relapse | Up to 12 months
  Time to early relapse of patients discharged from a short-stay psychiatric hospitalisation unit.
Number of readmission of patients | Up to 12 months
  Readmission in short-stay psychiatric hospital units when the schizophrenia or schizoaffective or schizophreniform disorder relapse.
Clinical Global Impression - Severity (CGI-S) Score | Up to 3 years
  The CGI-S rating scale is used to rate the severity of a patient's psychotic condition on a 7-point scale. It is rated as follows: 1=Normal, not at all ill, 2=Borderline mentally ill, 3=Mildly ill, 4=Moderately ill, 5=Markedly ill, 6=Severely ill, and 7=Among the most extremely ill. Higher scores indicate worsening.

SECONDARY OUTCOMES:
Duration of disease | Within 3 years before the study start
Drug abuse | Within 3 years before the study start
Psychiatric diagnosis | Within 3 years before the study start
  Patients diagnosed with Schizophrenia or Schizoaffective/schizophreniform disorder.
Previous stress or event | Within 3 years before the study start
Hospitalizations in the previous 3 years | Within 3 years before the study start
Adherence to the psychiatric treatment | Within 3 years before the study start
Previous pharmacological treatment | Within 3 years before the study start

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag S.A., Spain Clinical Trial, Study Director — Janssen-Cilag, S.A.

REFERENCES:
- See also: Scale Validation of Prediction of Relapse and Rehospitalization Short Term in Patients with Schizophrenia — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=286&filename=CR011989_CSR.pdf